CLINICAL TRIAL: NCT01788618
Title: Cancer and Disorders of Cognitive Functions and Quality of Life: "Cognitive Rehabilitation in Patients Suffering From Cancer and Treated With Chemotherapy"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Francois Baclesse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: COG REDUC
Record Dates: First submitted 2013-02-08; First posted 2013-02-11 (Estimated); Last update posted 2017-07-28 (Actual); Status verified 2015-08

CONDITIONS: Cancer
Keywords: Cognitive functions; Quality of life; Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Experimental group (Other): Cognitive exams at T0 and T3. Patients will achieve 9 standardized cognitive rehabilitation sessions with the RehaCom ® software (over 3 months), and a self-assessment of their monthly experienced cognitive functioning using the self-administered questionnaire FACT-Cog
  Interventions: Other: Cognitive exams; Other: standardized cognitive rehabilitation
- The control group 1 (Homework) (Other): Cognitive exams at T0 and T3. These patients will take part in 9 sessions standardized home exercise (over 3 months), and a self-assessment every month felt their cognitive functioning using the self-administered questionnaire FACT Cog
  Interventions: Other: Cognitive exams; Other: Standardized home exercise
- Control group 2 ( telephone follow) (Other): Cognitive exams at T0 and T3. These patients receive follow-up by phone (9 telephone calls over a period of 3 months) standardized optics to know the evolution of the disorder and felt the same way as for the other groups, a monthly self-assessment the feeling of cognitive functioning using the self-administered questionnaire FACT-Cog
  Interventions: Other: Cognitive exams; Other: Follow up by phone

INTERVENTIONS:
Other: Cognitive exams — Psychopathological assessment (T0 and T3):
  * Scale of Spielberger
  * The self-administered questionnaire CES-D
  Cognitive assessment(T0 and T3):
  - MMS, Grober and Buschke test, memory for numbers (WAIS IV) sequence of numbers and letters (WAIS IV), arithmetic (WAIS IV), Trail Making Test, verbal Fluence, D2, Code (WAIS IV)
  Quality of Life: FACT-G and FACT-An Fatigue Module (T0 and T3):
  Self-assessment FACT-COG (T0,every months until T3)
Other: standardized cognitive rehabilitation — Patients will achieve 9 standardized cognitive rehabilitation sessions with the RehaCom ® software (over 3 months), and a self-assessment of their monthly experienced cognitive functioning using the self-administered questionnaire FACT-Cog
  Arms: Experimental group
Other: Standardized home exercise — These patients will take part in 9 sessions standardized home exercise (over 3 months), and a self-assessment every month felt their cognitive functioning using the self-administered questionnaire FACT Cog
  Arms: The control group 1 (Homework)
Other: Follow up by phone — These patients receive follow-up by phone (9 telephone calls over a period of 3 months) standardized optics to know the evolution of the disorder and felt the same way as for the other groups, a monthly self-assessment the feeling of cognitive functioning using the self-administered questionnaire FACT-Cog
  Arms: Control group 2 ( telephone follow)

SUMMARY:
Our study aims to measure the impact of cognitive rehabilitation workshops on the development of cognitive functions and quality of life of patients expressing a cognitive complaint

DETAILED DESCRIPTION:
The main objective of our study was to evaluate, in patients treated for cancer expressing the cognitive complaint during or after treatment, interest workshops on improving cognitive rehabilitation felt their cognitive functions and their quality of life.

The primary endpoint was the proportion of patients showing an improvement in the score of perceived deficiencies (score ranging from 0 to 72) of the FACT-Cog after treatment. The FACT-Cog is a self-administered questionnaire assessing the patients felt their cognitive difficulties (memory, attention, concentration) and the impact of these difficulties on their quality of life. The improvement is defined as an increase of 7 points >= cognitive score won by the (a) patient (e) after the treatment

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years
* Solid tumor or haematological
* Chemotherapy and / or targeted therapy in the adjuvant or metastatic
* Sequential processing
* Subjective cognitive complaints during or after treatment assessed by four items of the FACT-COG (impact on quality of life). Score ≥ 4/16 questions Q35, Q37, Q38 and Q41 FACT COG - Patient in remission or pause therapeutic
* Subjective between 1 month and 5 years after the end of chemotherapy and / or targeted therapy cognitive complaints (ongoing treatment with Herceptin is not a non-inclusion criteria)
* Lack of personality disorders and / or psychiatric disorder scalable
* No known brain metastases
* Lack of primary brain tumor
* Lack of analgesic treatment with opioids or Class 3
* Having signed informed consent to participate in the study
* Mastery of the French language

Exclusion Criteria:

* Primary cancer of the central nervous system or brain metastases
* Pathology malignant hematologic
* Disorders of higher functions documented
* Pathology psychiatric scalable
* Use documented drug
* Cancer treated in childhood
* Patient or opioids analgesics in Class 3
* Consumption of alcohol
* Patient unable to respond to cognitive tests and cognitive rehabilitation
* Refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2012-07; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Proportion of patients showing an improvement in the score of perceived deficiencies (score ranging from 0 to 72) of the FACT-Cog after care | up to 3 months
  Evaluate, in patients treated for cancer expressing a cognitive complaint during or after the treatment, the interest workshops on improving cognitive rehabilitation felt their cognitive function and quality of life.
  Autoquestionnary FACT COG

SECONDARY OUTCOMES:
Evaluate the relationship between cognitive impairment and the parameters of the quality of life | Baseline and month 3
  Cognitive assessment:
  MMS, Test de Grober et Buschke, mémoire des chiffres (WAIS IV), séquence lettres-chiffres (WAIS IV), arithmétique (WAIS IV), Trail Making Test, Fluence verbale, D2, Code (WAIS IV)
Assess the relationships between goals disorders (measured by neuropsychological tests) and the patients felt | Baseline and month 3
  Cognitive assessment:
  MMS, Test de Grober et Buschke, mémoire des chiffres (WAIS IV), séquence lettres-chiffres (WAIS IV), arithmétique (WAIS IV), Trail Making Test, Fluence verbale, D2, Code (WAIS IV)
Study of different types of interest support the evolution of objective and subjective cognitive performance of patients | Baseline and month 3
  Cognitive assesment:
  MMS, Test de Grober et Buschke, mémoire des chiffres (WAIS IV), séquence lettres-chiffres (WAIS IV), arithmétique (WAIS IV), Trail Making Test, Fluence verbale, D2, Code (WAIS IV)

CONTACTS AND LOCATIONS:
Overall Officials: Florence JOLY-LOBBEDEZ, PHD, Principal Investigator — Centre François Baclesse
Locations (4):
- France (4):
  - Centre François Baclesse, Caen
  - Centre Henri Becquerel, Rouen
  - Centre Paul Strauss, Strasbourg
  - Institut Gustave Roussy, Villejuif